CLINICAL TRIAL: NCT03828032
Title: Alternations of Multi-parameters Including Hemodynamic Concentration and Water Levels During Dehydration Therapy on Brain Edema Patients
Brief Title: Multi-parameters'Change Process During Dehydration Therapy on Brain Edema Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ting Li (Unknown)
Collaborators: Affiliated Hospital of Armed Police Logistics College (Unknown)
Responsible Party: Sponsor-Investigator, Ting Li, Fellow, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Brain edema dehydration
Record Dates: First submitted 2019-01-31; First posted 2019-02-04 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Hemodynamic Instability; Water on the Brain; Intracranial Pressure Increase
Keywords: Brain edema; dehydration; Noninvasive optical method
MeSH Terms: conditions — Hydrocephalus; Intracranial Hypertension; Brain Edema; Dehydration | interventions — Mannitol; Saline Solution, Hypertonic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mannitol injection (Experimental): The participant receive mannitol injection to decrease intracranial pressure in the ward with optical probes on his/her forehead.
  Interventions: Procedure: Mannitol injection
- Hypertonic saline injection (Experimental): The participant receive hypertonic saline of specific concentration injection to decrease intracranial pressure in the ward with optical probes on his/her forehead.
  Interventions: Procedure: Hypertonic saline injection

INTERVENTIONS:
Procedure: Mannitol injection — Standard mannitol injection to decrease intracranial pressure of patients
  Arms: Mannitol injection
Procedure: Hypertonic saline injection — Standard Hypertonic saline injection to decrease intracranial pressure of patients
  Arms: Hypertonic saline injection

SUMMARY:
This study aims to investigate the inner mechanism during different dehydration therapies such as mannitol injection and hypertonic saline. The investigators used a self-made near infrared spectroscopy (NIRS) instrument to monitor the physiological changes noninvasively including oxyhemoglobin ([HbO2]), deoxy-hemoglobin ([Hb]), the derived change in blood volume ([tHb]) and water concentration on the forehead of brain edema patients.

DETAILED DESCRIPTION:
Cerebral edema, as an acute head injury along with high intracranial pressure, has been of great interest over decades in clinical neurosurgery research. Dehydration therapy is a common clinical method to decrease intracranial pressure. This study aims to investigate the inner mechanism during different dehydration therapies such as mannitol injection and hypertonic saline. The investigators used a self-made near infrared spectroscopy (NIRS) instrument to monitor the physiological changes noninvasively including oxyhemoglobin ([HbO2]), deoxy-hemoglobin ([Hb]), the derived change in blood volume ([tHb]) and water concentration on the forehead of brain edema patients. Then the investigators compared the changes process of multiple physiological parameters during different dehydration therapies.

ELIGIBILITY:
Inclusion Criteria:

• Patients who had brain edema and need dehydration therapy to decrease intracranial pressure.

Exclusion Criteria:

* AIDS, Active Hepatitis, Tuberculosis, Syphilis
* Patients who regularly take anticoagulants, antiplatelet drugs
* Anemia, thrombocytopenia
* Hemorrhagic disease like hemophilia

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-12-11 (Estimated)

PRIMARY OUTCOMES:
Δ[HbO2] | 2 weeks
  changes of oxyhemoglobin concentration
water concentration | 2 weeks
  water concentration of brain

SECONDARY OUTCOMES:
intracranial pressure | 2 weeks
  intracranial pressure
Δ[Hb] | 2 weeks
  changes of deoxy-hemoglobin concentration

IPD SHARING:
Plan to Share IPD: No